CLINICAL TRIAL: NCT03937258
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO ASSESS SINGLE DOSE AND MULTIPLE DOSE PHARMACOKINETICS OF PF-04965842 AND ITS METABOLITES, AND THE EFFECT OF REPEAT-DOSE PROBENECID ON THE SINGLE DOSE PHARMACOKINETICS OF PF-04965842 AND ITS METABOLITES IN HEALTHY PARTICIPANTS
Brief Title: A Study to Assess Pharmacokinetics of PF-04965842 and Its Metabolites and Effect of Probenecid in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: B7451043
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — abrocitinib; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-04965842 single dose (Other): In Period 1, subjects will be administered a single oral 200 mg dose of PF 04965842 in the morning on Day 1 under fasted conditions.
  Interventions: Drug: PF-04965842
- PF-04965842 multiple doses (Other): In Period 2, participants will receive oral 200 mg dose of PF-04965842 once daily (QD) in the morning of Day 1 to Day 4 under fasted conditions.
  Interventions: Drug: PF-04965842
- Probenecid and PF-04965842 (Other): In Period 3, participants will receive probenecid 1000 mg twice daily (BID) in the mornings and evenings of Day 1 to Day 3. On the morning of Period 3 Day 2, after an overnight fast of approximately 8 hours, participants will be administered probenecid 1000 mg. A single 200 mg oral dose of PF 04965842 will be administered approximately 2 hours after the probenecid dose.
  Interventions: Drug: PF-04965842; Drug: Probenecid

INTERVENTIONS:
Drug: PF-04965842 — Participants will be administered a single oral 200 mg dose of PF-04965842 in the morning on Period 1 Day 1 and Period 3 Day 2 under fasted conditions. In Period 2, participants will receive oral 200 mg dose of PF-04965842 once daily (QD) in the morning of Day 1 to Day 4 under fasted conditions
Drug: Probenecid — In Period 3, participants will receive probenecid 1000 mg twice daily (BID) in the mornings and evenings of Day 1 to Day 3. On the morning of Period 3 Day 2, after an overnight fast of approximately 8 hours, participants will be administered probenecid 1000 mg. A single 200 mg oral dose of PF 04965842 will be administered approximately 2 hours after the probenecid dose.
  Arms: Probenecid and PF-04965842

SUMMARY:
A total of approximately 12 healthy male or female participants will be enrolled in the study so that at least 10 participants will complete the study.

Participants will be screened within 28 days of the first dose of study medication. The single fixed-sequence will consist of 3 periods. Participants will report to the clinical research unit (CRU) at least 12 hours prior to Day 1 dosing in Period 1 and will be required to stay in the CRU for 12 days and 11 nights. Genotyping samples for cytochrome P450 (CYP) 2C19 and CYP2C9 will be collected pre dose in Period 1 only.

In Period 1, participants will be administered a single oral 200 mg dose of PF-04965842 in the morning on Day 1 under fasted conditions (overnight fasting for at least 10 hours). No food will be allowed for at least 4 hours postdose and undergo serial blood sample collection for 48 hours postdose.

In Period 2, participants will receive oral 200 mg dose of PF-04965842 once daily (QD) in the morning of Day 1 to Day 4 under fasted conditions (overnight fasting for at least 10 hours). No food will be allowed for at least 4 hours postdose and undergo serial blood sample collection for 48 hours postdose on Day 4.

In Period 3, participants will receive probenecid 1000 mg twice daily (BID) in the mornings and evenings of Day 1 to Day 3. On the morning of Period 3 Day 2, after an overnight fast of approximately 8 hours, participants will be administered probenecid 1000 mg. A single 200 mg oral dose of PF 04965842 will be administered approximately 2 hours after the probenecid dose. Participants will remain in a fasted state for 4 hours after dosing with PF 04965842 and undergo serial blood sample collection for 48 hours post PF 04965842 dosing. Participants will be discharged from the CRU on Day 4 after all study procedures are completed. The participant will be required to have a Follow-up phone contact 28-35 days after the last dose of investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female participants who are overtly healthy as determined by medical evaluation including detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12-lead ECG, and clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent , which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing). Evidence of acute exacerbation of dermatological condition (eg, AD, eczema or psoriasis) or visible rash present during physical examination. Participants with history of psoriasis, AD or eczema can be included in the study.
2. Participants, who according to the product label for probenecid, would be at increased risk if dosed with probenecid, including participants with known blood dyscrasias, uric acid kidney stones, gout, or gouty arthritis.
3. Any condition possibly affecting drug absorption (eg, gastrectomy).
4. Known relevant history or current elevations of liver function tests (LFTs) or impaired liver function.
5. History of active or latent or inadequately treated tuberculosis (TB) infection, or a positive QuantiFERON- TB Gold test.
6. Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of screening. History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized multi-dermatomal herpes zoster.
7. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C virus antibody (HCVAb). Hepatitis B vaccination is allowed.
8. History or evidence of any malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
9. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
10. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
11. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
12. A positive urine drug test.
13. Screening supine systolic blood pressure (BP) <= 140 mm Hg or <90 mm Hg, following at least 5 minutes of supine rest OR Screening supine diastolic BP <50 mm Hg or >= 90 mm Hg following at least 5 minutes of supine rest. If a participant meets any of these criteria, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
14. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility.
15. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    1. Absolute neutrophil count of <1200/mm3;
    2. Hemoglobin <10.0 g/dL or hematocrit <30%;
    3. Absolute lymphocyte count <500/mm3;
    4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level>= 2 * upper limit of normal (ULN);
    5. Total bilirubin level >1 * ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN;
    6. Uric acid not within the normal reference range;
    7. Platelet count of <150,000/mm3;
    8. Estimated creatinine clearance <40 mL/min based on the age appropriate calculation, or serum creatine >1.5 times the ULN.
16. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
17. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or 2 chews of tobacco per day.
18. Pregnant female participants; breastfeeding female participants; female participants of childbearing potential who are unwilling or unable to use 1 highly effective method of contraception as outlined in this protocol Contraception section for the duration of the study and for at least 28 days after the last dose of investigational product.
19. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
20. History of sensitivity to heparin or heparin-induced thrombocytopenia.
21. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
22. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of PF-04965842 | Period 1 Day 1, and Period 3 Day 2.
Area under the curve from time zero to extrapolated infinite time (AUCinf) of PF-04965842 | Period 1 Day 1 and Period 3 Day 2
AUC from time 0 to the time of the last quantifiable concentration (AUClast) of PF-04965842 | Period 1 Day 1 and Period 3 Day 2
Area under the plasma concentration-time profile from time 0-24hr (AUCtau) of PF-04965842 | Period 1 Day 1

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs). | Screening up to 28-35 days after the last dose of PF 04965842 in period 3
  Number of subjects with adverse events (AEs).
Number of subjects with laboratory tests findings of potential clinical importance | Screening up to Period 3 Day 4
  Number of subjects with laboratory tests findings of potential clinical importance
Number of subjects with clinically significant abnormal vital signs | Screenig up to Period 3 Day 4
  Number of subjects with clinically significant abnormal vital signs
Number of subjects with clinically significant abnormal Electrocardiograms (ECGs) | Screening up to Period 3 Day 4
  Number of subjects with clinically significant abnormal Electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Wouters A, Tatulych S, Connell CA, Le VH, Tripathy S, O'Gorman MT, Winton JA, Yin N, Valdez H, Malhotra BK. Assessment of the Effects of Inhibition or Induction of CYP2C19 and CYP2C9 Enzymes, or Inhibition of OAT3, on the Pharmacokinetics of Abrocitinib and Its Metabolites in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2022 May;47(3):419-429. doi: 10.1007/s13318-021-00745-6. Epub 2022 Feb 28. PMID 35226304
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451043